CLINICAL TRIAL: NCT03832907
Title: Inpatient and Post-hospital Discharge Assessment of Glycemic Control by Capillary Point-of-care Glucose Testing and by Continuous Glucose Monitoring in Insulin-treated Patients With Type 1 and Type 2 Diabetes: Dexcom G6 Observational Study
Brief Title: Dexcom G6 Observational Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00107627
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Diabetes
Keywords: Glucose monitoring; POC BG; DexcomG6 CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dexcom G6 CGM - Continues Glucose Monitoring sensor system (Experimental): The Dexcom G6 CGM is a commercially available factory-calibrated sensor system. The system measures interstitial glucose every 5-15 minutes, providing real-time and more complete glycemic profile during 24-hours compared to standard POC glucose testing, and replaces the need for finger sticking. Potential limitations include the need for removing the sensor before MRI or diathermy treatment, and the potential interference in patients with severe dehydration.
  In parallel, same participants will be monitored by the standard of care point-of-care (POC) capillary glucose tests. Diabetes guidelines recommend bedside capillary POC testing before meals and at bedtime to assess glycemic control and to adjust insulin therapy in the hospital.
  Interventions: Device: Dexcom G6 CGM - Continues Glucose Monitoring sensor system; Diagnostic Test: POC BG - Point-of-Care Blood Glucose monitoring

INTERVENTIONS:
Device: Dexcom G6 CGM - Continues Glucose Monitoring sensor system — A blinded factory-calibrated continues glucose monitoring sensor system Dexcom G6 will be placed shortly after admission. Two CGM devices will be inserted in all patients - one in the abdomen and one in the arm to also assess differences in blood glucose readings between upper extremity and abdominal insertion sites. Information on CGM readings will be collected daily during the hospital stay and after hospital discharge for 10 days using the Dexcom Studio software to download the Dexcom receiver data.
Diagnostic Test: POC BG - Point-of-Care Blood Glucose monitoring — Standard of care - bedside point-of-care (POC) capillary blood glucose (BG) monitoring will be done before meals and bedtime daily during the hospital stay and after hospital discharge for 10 days.
  Other Names: Standard of Care capillary glucose test

SUMMARY:
This is an exploratory prospective study primary aiming to evaluate differences between Point-of-care (POC) testing (standard of care) and Dexcom G6 CGM (Continues Glucose Monitoring sensor system) in 1) glycemic control measured by mean daily blood glucose and 2) identifying hypoglycemic and hyperglycemic events - in patients with type 1 and type 2 diabetes treated with basal bolus insulin regimen.

DETAILED DESCRIPTION:
Several studies have shown that the use of a device that can measure blood glucose levels every 5 minutes is more effective in identifying low blood glucose (hypoglycemia) and high blood glucose (hyperglycemia) when compared to regular measurements with fingersticks [point of care (POC)].

This is an exploratory prospective study primary aiming to evaluate differences between Point-of-care (POC) testing (standard of care) and Dexcom G6 CGM (Continues Glucose Monitoring sensor system) in 1) glycemic control measured by mean daily blood glucose and 2) identifying hypoglycemic and hyperglycemic events - in patients with type 1 and type 2 diabetes treated with basal bolus insulin regimen.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years admitted to a general medicine or surgical service.
2. Known history of T1D or T2D receiving insulin therapy
3. Subjects must have a randomization BG between 140 mg and 400 mg/dL without laboratory evidence of diabetic ketoacidosis (bicarbonate < 18 mEq/L, pH < 7.30, or positive serum or urinary ketones).
4. Patients with expected hospital length-of-stay of 3 or more days

Exclusion Criteria:

1. Patients with acute illness admitted to the ICU or expected to require admission to the ICU.
2. Patients expected to require MRI procedures during hospitalization.
3. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
4. Female subjects who are pregnant or breast-feeding at time of enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Started | 101
Completed | 91
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 85
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose by POC Reading сompared to CGM Reading
Description: Mean daily blood glucose will be calculated
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
mg/dL
  POC | 175.55 (42.37)
  CGM | 175.84 (42.35)

2. Primary Outcome: Number of Clinical Significant Hypoglycemia (<54 mg/dl) Events by POC Reading Compared to CGM Reading
Description: Number of clinical significant hypoglycemia (<54 mg/dl) events will be calculated
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 9
  CGM | 60

3. Primary Outcome: Number of Severe Hyperglycemia (>240 mg/dl) Events by POC Reading Compared to CGM Reading
Description: Number of severe hyperglycemia (>240 mg/dl) events will be recorded
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 305
  CGM | 518

4. Secondary Outcome: Mean Daily Blood Glucose by POC Reading Compared to CGM Reading
Description: Mean daily blood glucose will be calculated
Time Frame: 10 days post discharge
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
mg/dL
  POC | 175.55 (42.37)
  CGM | 173.13 (41.77)

5. Secondary Outcome: Number of Clinical Significant Hypoglycemia (<54 mg/dl) Events by POC Reading Compared to CGM Reading
Description: Number of clinical significant hypoglycemia (<54 mg/dl) events will be calculated
Time Frame: 10 days post discharge
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 9
  CGM (arm) | 29

6. Secondary Outcome: Number of Clinical Significant Severe Hyperglycemia (>240 mg/dl) Events by POC Reading Compared to CGM Reading
Description: Number of severe hyperglycemia (>240 mg/dl) events will be recorded
Time Frame: 10 days post discharge
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 305
  CGM | 399

7. Secondary Outcome: Number of Nocturnal Hypoglycemic Events < 70 mg/dl (Between 22:00 and 06:00) by POC Reading Compared to CGM Reading
Description: Number of nocturnal hypoglycemic events < 70 mg/dl (between 22:00 and 06:00) will be recorded
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 1
  CGM abdomen | 48
  CGM arm | 34

8. Secondary Outcome: Number of Nocturnal Hypoglycemic Events < 70 mg/dl (Between 22:00 and 06:00) by POC Reading Compared to CGM Reading
Description: Number of nocturnal hypoglycemic events < 70 mg/dl(between 22:00 and 06:00) will be recorded
Time Frame: 10 days post discharge
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 1
  CGM abdomen | 22
  CGM arm | 9

9. Secondary Outcome: Number of of Hypoglycemic Events < 70mg/dl in POC Group by POC Reading Compared to CGM Reading
Description: Number of of hypoglycemic events < 70mg/dl will be recorded
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 36
  CGM abdomen | 144
  CGM arm | 115

10. Secondary Outcome: Number of Hypoglycemic Events < 70mg/dl by POC Reading Compared to CGM Reading
Description: Number of of hypoglycemic events < 70mg/dl will be recorded
Time Frame: 10 days post discharge
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 10
  CGM abdomen | 100
  CGM arm | 48

11. Secondary Outcome: Time in Hypoglycemia (Minutes) During the Day and Night by CGM Reading
Description: Time in hypoglycemia (minutes) during the day and night will be recorded. Only measured by CGM, Discrete POC values are not used to assess amount of time spent within a specific glucose range. .
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
min
  CGM abdomen) | 119.08 (216.56)
  CGM arm | 78.63 (135.33)

12. Secondary Outcome: Time in Hypoglycemia (Minutes) During the Day and Night by CGM Reading
Description: as for outcome 11
Time Frame: 10 days post discharge
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
min
  CGM abdomen | 118.70 (217.83)
  CGM arm | 89.14 (140.16)

13. Secondary Outcome: Time in Hyperglycemia (Minutes) During the Day and Night> 240 mg/dl by CGM Reading
Description: Time in hyperglycemia (minutes) during the day and night> 240 mg/dl will be recorded. Only measured by CGM, Discrete POC values are not used to assess amount of time spent within a specific glucose range. .
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
min
  CGM abdomen | 972.30 (1214.5)
  CGM arm | 723.23 (1061.4)

14. Secondary Outcome: Time in Hyperglycemia (Minutes) During the Day and Night> 240 mg/dl by CGM Reading
Description: Time in hyperglycemia (minutes) during the day and night> 240 mg/dl will be recorded. Only measured by CGM, Discrete POC values are not used to assess amount of time spent within a specific glucose range.
Time Frame: 10 days post discharge
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
min
  CGM abdomen | 4624.3 (13554)
  CGM arm | 1706.1 (2255.6)

15. Secondary Outcome: Number of Hyperglycemic Events > 240 mg/dl by POC Reading Compared to CGM Reading
Description: Number of hyperglycemic events > 240 mg/dl will be recorded
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 305
  CGM abdomen | 518
  CGM arm | 399

16. Secondary Outcome: Number of Hyperglycemic Events > 240 mg/dl by POC Reading Compared to CGM Reading
Description: Number of hyperglycemic events > 240 mg/dl will be recorded
Time Frame: 10 days post discharge
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 153
  CGM abdomen | 554
  CGM arm | 316

17. Secondary Outcome: Percentage of BG Readings Within Target BG of 70 and 180 mg/dl by POC Reading Compared to CGM Reading
Description: Percentage of BG readings within target BG of 70 and 180 mg/dl will be calculated
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Mean (Standard Deviation); unit: percentage of readings
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of readings
  POC | 59.70 (24.73)
  CGM (abdomen) | 58.91 (26.83)
  CGM arm | 60.97 (28.56)

18. Secondary Outcome: Percentage of BG Readings Within Target BG of 70 and 180 mg/dl by POC Reading Compared to CGM Reading
Description: Percentage of BG readings within target BG of 70 and 180 mg/dl will be calculated
Time Frame: 10 days post discharge
Measure: Mean (Standard Deviation); unit: percentage of readings
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of readings
  POC | 59.56 (29.31)
  CGM abdomen | 52.62 (30.64)
  CGM arm | 51.60 (31.94)

19. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Below Glucose Target <70mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time below glucose target <70mg/dl will be calculated. Only measured by CGM, Discrete POC values are not used to assess amount of time spent within a specific glucose range.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of readings
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of readings
  CGM <70 abdomen | 10
  CGM <70 arm | 4.6

20. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Below Glucose Target <70 mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time below glucose target <70 mg/dl will be calculated
Time Frame: 10 days post discharge
Measure: Number; unit: percentage of patients
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of patients
  CGM abdomen | 5.3
  CGM arm | 2.9

21. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Above Glucose Target >180mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time above glucose target >180 mg/dl will be calculated
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of patients
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of patients
  CGM abdomen | 91
  CGM arm | 89

22. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Above Glucose Target >180 mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time above glucose target >180 will be calculated
Time Frame: 10 days post discharge
Measure: Number; unit: percentage of patients
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of patients
  CGM abdomen | 89
  CGM arm | 94

23. Secondary Outcome: Glycemic Variability Calculated by Standard Deviation by CGM Reading
Description: Glycemic variability will be calculated using Standard Deviation
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
mg/dl
  CGM abdomen | 46.37 (15.45)
  CGM arm | 43.37 (15.31)

24. Secondary Outcome: Glycemic Variability Calculated by MAGE by CGM Reading
Description: MAGE: average amplitude of glycemic excursions with values exceeding a certain threshold.
Time Frame: 10 days post discharge
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
mg/dl
  CGM abdomen | 58.33 (24.43)
  CGM arm | 55 (23.76)

25. Secondary Outcome: Number of Sensor Removal/Failures/Dislodgments
Description: Number of sensor removal/failures/dislodgments will be recorded
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events | 31

26. Secondary Outcome: Mean Absolute Relative Difference (MARD) of CGM Compared to POC
Description: Accuracy of Dexcom G6 CGM, as defined by overall MARD, compared to POC
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Mean (Standard Deviation); unit: percent difference
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percent difference
  CGM abdomen | 12.54 (15.24)
  CGM arm | 12.22 (15.11)

27. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 30/30% for Values < 70 mg/d Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values in the hypoglycemic range (<70 mg/dl) meeting %30/30 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 89.3
  CGM arm | 85.2

28. Secondary Outcome: Percentage of Values Within Zone A, B, C, D of the Clarke Error Grid Measured in Abdomen
Description: Percentage of CGM glucose values within defined performance zones (A-E) indicating potential for clinical error. The Clarke error grid analysis uses a Cartesian diagram, in which the estimated/predicted values are displayed on the y-axis, whereas the reference values are presented on the x-axis. This diagram is subdivided into 5 zones: A, B, C, D, and E. The points that fall within zones A and B represent, respectively, sufficiently accurate and acceptable glucose results (better outcome), points in zone C may prompt unnecessary corrections, points in zones D and E represent erroneous and incorrect treatment.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  A | 82.4
  B | 16.5
  C | 0.1
  D | 1

29. Secondary Outcome: Percentage of Values Within Zone A, B, C of the Clarke Error Grid Measured in Arm
Description: as for outcome 28
Time Frame: During hospital stay (3 days - up to 30 days) measured in arm
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  A | 81.4
  B | 17.6
  C | 0.1
  D | 0.9

30. Secondary Outcome: Number of Nocturnal Hypoglycemic Events < 54 mg/dl (Between 22:00 and 06:00) by POC Reading Compared to CGM Reading
Description: Number of nocturnal hypoglycemic events < 54 mg/dl (between 22:00 and 06:00) will be recorded
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 1
  CGM abdomen | 12
  CGM arm | 4

31. Secondary Outcome: Number of Nocturnal Hypoglycemic Events < 54 mg/dl (Between 22:00 and 06:00) by POC Reading Compared to CGM Reading
Description: Number of nocturnal hypoglycemic events < 54 mg/dl(between 22:00 and 06:00) will be recorded
Time Frame: 10 days post discharge
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 0
  CGM abdomen | 8
  CGM arm | 3

32. Secondary Outcome: Number of of Hypoglycemic Events < 54 in POC Group by POC Reading Compared to CGM Reading
Description: Number of of hypoglycemic events < 54 will be recorded
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 9
  CGM abdomen | 60
  CGM arm | 29

33. Secondary Outcome: Number of Hypoglycemic Events < 54mg/dl by POC Reading Compared to CGM Reading
Description: Number of of hypoglycemic events < 54mg/dl will be recorded
Time Frame: 10 days post discharge
Measure: Number; unit: number of events
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
number of events
  POC | 3
  CGM abdomen | 48
  CGM arm | 16

34. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Below Glucose Target <54mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time below glucose target <54mg/dl will be calculated. Only measured by CGM, Discrete POC values are not used to assess amount of time spent within a specific glucose range.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of patients
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of patients
  CGM <70 abdomen | 3.4
  CGM <70 arm | 0

35. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Above Glucose Target >240 mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time above glucose target >240 will be calculated
Time Frame: 10 days post discharge
Measure: Number; unit: percentage of patients
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of patients
  CGM abdomen | 56
  CGM arm | 60

36. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Above Glucose Target >240 mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time above glucose target >240 mg/dl will be calculated
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of patients
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of patients
  CGM abdomen | 53
  CGM arm | 43

37. Secondary Outcome: Glycemic Variability Calculated by MAGE by CGM Reading
Description: The average amplitude of glycemic excursions with values exceeding a certain threshold.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
mg/dl
  CGM abdomen | 58.73 (27.87)
  CGM arm | 56.68 (30.87)

38. Secondary Outcome: Percentage of Patients With Greater Than 5%-Time Below Glucose Target <54 mg/dl by CGM Reading
Description: Percentage of patients with greater than 5%-time below glucose target <54 mg/dl will be calculated
Time Frame: 10 days post discharge
Measure: Number; unit: percentage of patients
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of patients
  CGM abdomen | 1.8
  CGM arm | 2.9

39. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 30/30% for Values 70-140 mg/dl Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values within the 70-140 mg/dl range that meet %30/30 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 93.1
  CGM arm | 92.9

40. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 30/30% for Values 140-180 mg/dl , Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values within the 140-180 mg/dl range that meet %30/30 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 93.3
  CGM arm | 94.9

41. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 30/30%for Values > 180 mg/dl, Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values in the hyperglycemic range (>180 mg/dl) that meet %30/30 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 95.5
  CGM arm | 94

42. Secondary Outcome: Glycemic Variability Calculated by Standard Deviation by CGM Reading
Description: Glycemic variability will be calculated using Standard Deviation
Time Frame: 10 days post discharge
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
mg/dl
  CGM abdomen | 46.37 (18.17)
  CGM arm | 43.87 (20.01)

43. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 20/20% for Values < 70 mg/dl Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values in the hypoglycemic range (<70 mg/dl) that meet %20/20 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 78.6
  CGM arm | 74.1

44. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 20/20% for Values 70-140 mg/dl Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values within the 70-140 mg/dl range that meet %20/20 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 82.0
  CGM arm | 82.0

45. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 20/20%for Values > 180 mg/dl, Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values in the hyperglycemic range (>180 mg/dl) that meet %20/20 accuracy criteria..
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 84.7
  CGM arm | 81.1

46. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 20/20% for Values 140-180 mg/dl , Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values within the 140-180 mg/dl range that meet %20/20 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 83.2
  CGM arm | 83.6

47. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 15/15% for Values < 70 mg/dl Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values in the hypoglycemic range (<70 mg/dl) that meet %15/15 accuracy criteria..
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 75.0
  CGM arm | 66.7

48. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 15/15% for Values 70-140 mg/dl Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values within the 70-140 mg/dl range that meet %15/15 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 69.4
  CGM arm | 70.5

49. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 15/15% for Values 140-180 mg/dl , Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values within the 140-180 mg/dl range that meet %15/15 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 69.6
  CGM arm | 73.8

50. Secondary Outcome: Percentage of Dexcom G6 CGM Sensor Values Within 15/15%for Values > 180 mg/dl, Compared to the Standard-of-care POC BG
Description: Percentage of CGM glucose values in the hyperglycemic range (>180 mg/dl) that meet %15/15 accuracy criteria.
Time Frame: During hospital stay (3 days - up to 30 days)
Measure: Number; unit: percentage of values
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
Number analyzed (Participants) | 91
percentage of values
  CGM abdomen | 71.0
  CGM arm | 71.5

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 4/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexcom G6 CGM - Continues Glucose Monitoring Sensor System (N=101)
Sensor site irritation/bleeding (Injury, poisoning and procedural complications) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT03832907/Prot_SAP_000.pdf